CLINICAL TRIAL: NCT00621439
Title: Exploratory Trial of Interferon Alpha-2b in Neoadjuvant Treatment of Ocular Melanoma
Brief Title: Investigative Trial of Interferon Alpha-2b To Shrink Cancer of the Eye
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding- study never began
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hans Grossniklaus, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00002566
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Ocular Melanoma
Keywords: ocular melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Receives 1 dose of Pegylated Interferon
  Interventions: Drug: Pegylated Interfon Alpha 2B
- II (Placebo Comparator): Receives placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pegylated Interfon Alpha 2B — Patients will receive PEG-IFN 6 mcg/kg subcutaneously 4 days prior to surgery. Patients will be premedicated with acetaminophen 700 mb orally prior to the injection. Only one dose of drug will be given. Enucleation will follow in 4 days.
  Arms: I
Drug: Placebo — Patients will receive placebo.
  Arms: II

SUMMARY:
The purpose of this study is to explore whether the drug pegylated-interferon-alfa-2b (PEG-IFN) has any effect on a certain type of immune cell (called natural killer cells) in patients with eye melanoma.

DETAILED DESCRIPTION:
The purpose of this study is to explore whether the drug pegylated-interferon-alfa-2b (PEG-IFN)has any effect on a certain type of immune cell (called natural killer cells) in patients with eye melanoma. Because this drug is currently being investigated for use against skin melanoma, we think this drug might have some benefit in eye melanoma as well, and that natural killer cells might be important in how the drug works.

Patients who choose to take part in the study will be randomized to receive either no drug, or PEG-IFN. Four days prior to the patient's surgery to remove the eye, 50cc of blood will be drawn. Patients who are randomized to PEG-IFN will be given the drug once, 4 days prior to surgery. Blood will also be drawn on the day of surgery (50cc), 1 week after surgery (50cc), 1 month (500cc), and 6 months (50cc).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have uveal melanoma for which enucleation is indicated, usually lesions greater than 8 mm in diameter and greater than 2 mm in thickness.
* Patients should have no evidence of metastatic disease as determined by history, physical examination, and appropriate liver injury enzymes.
* Patients should have received no prior interferon.
* Age >18 years.

Because of limited data on the use of pegylated interferon in patients <18 years of age and uncertainties about possible differences in NK response, children are excluded from this study. Since ocular melanoma is rare in children this is not expected to be an issue.

* Life expectancy of greater than 3 months
* ECOG performance status of 0- 2 (Karnofsky 60% or better; see Appendix II).
* Patients must have normal organ and marrow function as defined below:
* Hgb >/= 12.5 g/dl or hematocrit >/= 38%

  * Leukocytes >3,000/mcL
  * Absolute neutrophil count >1,500/mcL
  * Platelets>100,000/mcL
  * Total bilirubin within normal institutional limits unless patient has Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) within normal institutional limits. Patients with elevated levels of either of these enzymes may be accepted if the elevations are less than or equal to 2x the institutional upper limit of normal and patient has a normal liver on CT or MRI.
  * Creatinine within normal institutional limits OR Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for one year after the study drug is given. Should a woman become pregnant or suspect she is pregnant while participating in this study,she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients who have had agents known to be immunosuppressive (e.g, glucocorticoids) within the 4 weeks prior to planned receipt of study drug.
* Patients receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because interferon alpha has the potential for teratogenic effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with interferon, breastfeeding should be discontinued if the mother is treated with this agent.
* HIV-positive patients are ineligible because of the known immunosuppression associated with this disease.
* Patients with history of other malignancies are eligible provided that they are clinically free of metastases at the time of the study.
* Patients who have donated blood in the 56 days prior to the 500cc blood draw in this study are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Evidence of anti-melanoma natural killer cell boost | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Grossniklaus, MD, Principal Investigator — Emory University